CLINICAL TRIAL: NCT04039126
Title: Comparison of the Effectiveness of Povidone-Iodine Alone to Povidone-Iodine-Tetracycline Combination for Chemical Pleurodesis in Malignant Pleural Effusion
Brief Title: Comparison of the Effectiveness of Povidone-Iodine Alone to Povidone-Iodine-Tetracycline Combination
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Hospital, Ibadan (Other)
Collaborators: West African College of Surgeons (Other)
Responsible Party: Principal Investigator, Dr. Jibril Khalil, Principal Investigator, University College Hospital, Ibadan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UI/EC/19/0177
Record Dates: First submitted 2019-07-27; First posted 2019-07-31 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Malignant Pleural Effusion
Keywords: MALIGNANT PLEURAL EFFUSSION
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Pleurodesis; Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: DOUBLE BLINDED, PARTIPANT ASIIGNED USING WINPEPI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATIENTS WITH MALIGNANT PLEURAL EFFUSION (Experimental): PARTICIPANTS WITH MALIGNANT PLEURAL EFFUSIONS REQUIRING PLEURODESIS, COMBINATION OD POVIDONE IODOONE-TETRCYCLINE TO BE USED.
  Interventions: Drug: CHEMICAL PLEURODESIS WITH POVIDONE-IODINE-TETRACYCLINE COMBINATION; Drug: CHEMICAL PLEURODESIS WITH POVIDONE-IODINE ALONE
- PATEINT WITH MALIGANT PLEURAL EFFUSION REQUIRNG PLEURODESIS (Active Comparator): TO USE POVIDONE IODINE ALONE IN THIS GROUP
  Interventions: Drug: CHEMICAL PLEURODESIS WITH POVIDONE-IODINE ALONE

INTERVENTIONS:
Drug: CHEMICAL PLEURODESIS WITH POVIDONE-IODINE-TETRACYCLINE COMBINATION — Pleurodesis is the obliteration of the pleural cavity by inducing adhesions of the visceral and parietal pleural layers, mostly used in patients with pleural effusions, pneumothorax (18). The use of pleurodesis to induce pleural symphysis between the pleural layers dates backs to the beginning of the 20th century by Benthune(19) and has continued to evolve with different Thoracic surgeons and researchers still looking for the ideal pleurodesis agent.
  Other Names: PLEURODESIS
  Arms: PATIENTS WITH MALIGNANT PLEURAL EFFUSION
Drug: CHEMICAL PLEURODESIS WITH POVIDONE-IODINE ALONE — 20mls of 10% povidone-iodine (Wosan Solution Povidone-Iodine Usp 10%, Jawa International Limited) is mixed with 10mls of 1% xylocaine and 30mls of water for injection added to the mixture, making also a total volume of 60mls of the the single pleurodesis agents alone, which will be instilled into the pleural space via the closed thoracotomy tube.
  Other Names: PLEURODESE

SUMMARY:
Title of study: Comparison of the Effectiveness of Povidone-Iodine alone to Povidone-Iodine--Tetracycline Combination for Chemical Pleurodesis in Malignant Pleural Effusion.

Research design: Prospective Randomized Controlled Clinical Trial. Background: Malignant pleural effusion (MPE) is commonly encountered in clinical practice among patients with malignancy. In addition to its association with major morbidities, it also poses a high risk of recurrence following drainage. Chemical pleurodesis is often required to achieve pleural adhesion and obliteration of the pleural space to prevent such recurrence. Several agents are in common use for chemical pleurodesis with mixed effectiveness.

DETAILED DESCRIPTION:
STRUCTURED SUMMARY Title of study: Comparison of the Effectiveness of Povidone-Iodine alone to Povidone-Iodine--Tetracycline Combination for Chemical Pleurodesis in Malignant Pleural Effusion.

Research design: Prospective Randomized Controlled Clinical Trial. Background: Malignant pleural effusion (MPE) is commonly encountered in clinical practice among patients with malignancy. In addition to its association with major morbidities, it also poses a high risk of recurrence following drainage. Chemical pleurodesis is often required to achieve pleural adhesion and obliteration of the pleural space to prevent such recurrence. Several agents are in common use for chemical pleurodesis with mixed effectiveness.

Methodology: 62 consenting but blinded patients with clinical features of MPE who are undergoing pleural drainage and have fulfilled the criteria for chemical pleurodesis will be grouped by block balanced randomization into two equal groups- A and B. All the patients in Group A (Test) will have pleurodesis done with a solution combining 1 gram of sterile Tetracycline powder with 20mls of 10% Povidone-iodinemixed with 10mls of 1% xylocaine (for local intrapleural anesthesia) and 30mls of sterile water for injection instilled through the chest tube into the pleural space, while allpatients in Group B (Active control) will have 20mls of 10% Povidone-iodine mixed with 10mls of 1% xylocaine and 30mls of sterile water for injection. Drainage and radiographic parameters will be collected prior to chest tube removal and during outpatient follow-up to assess the effectiveness of pleurodesis in each group.

Objectives: To determine if combining tetracycline with 10% Povidone-iodine increases its effectiveness in pleurodesis for MPE.

Principal Exposure:Chemical pleurodesis with 10% Povidone-Iodine or combination of 10% Povidone-iodine-Tetracycline (1 gram).

Outcome variables: The primary outcome variable is the success of the pleurodesis in controlling MPE at 1month and 3 months follow-up. Success of pleurodesis classified as been Complete pleurosesis or Failed pleurodesis. The secondary outcome variables are: post-procedure complications of pain, hypotension,fever and occurrence of empyema thoracis, duration of thoracostomy tube retention post-pleurodesis, need for repeat of the procedure Keywords: Malignant Pleural Effusion, Chemical Pleurodesis, 10% Povidone-iodine, Tetracycline, Effectiveness

ELIGIBILITY:
Inclusion Criteria:

* • All adult patients aged between18- 70 years presenting with pleural effusion in association with a malignant disease.

  * Patients with documented malignant pleural effusion ( i.e positive pleural fluid for malignant cells on pleural fluid cytology and/or positive pleural biopsy for malignant tissue).
  * Reaccumulation of an effusion after drainage or patients presenting with symptoms related to pleural fluid re-accumulation such as dyspnea, cough and chest pain.
  * Patient with full lung re-expansion after thoracostomy tube insertion and drainage of effusion.

Exclusion Criteria:

* • Patients with known hypersensitivity either to Povidone-iodine and/or Tetracycline

  * Failure to achieve full lung re-expansion following drainage of the effusion within 48hrs
  * Locoregional radiotherapy to the effusion side.
  * Loculated pleural effusion
  * Refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Success of pleurodesis | 1 AND 3 MONTH AFTER PLEURODESIS
  classified as either a Complete Pleurodesis or Failed Pleurodesis. Complete pleurodesis defined as absence of pleural fluid re-accumulation on a chest radiograph at 1 and 3 months post-chemical pleurodesis, while Failed pleurodesis defined as pleural fluid re-accumulation requiring additional tube thoracostomy drainage before or at 1- 3 month follow up.

SECONDARY OUTCOMES:
Adverse Effects from the chemical pleurodesis agent used | immediate post procedure( 30minutes and 1 hour)
  Adverse effects which are Post-procedure Pain, Hypotension, Fever and development of Empyema Thoracis following pleurodesis.

CONTACTS AND LOCATIONS:
Overall Officials: catherine Falade, Prof., Study Chair — institute for advanced medical research and training, UI, IBADAN
Locations (1):
- University College Hospital,, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
proforma of the study, with theinformation gathered during the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: as the study is being conducted
Access Criteria: via email

REFERENCES:
- [Background] Psallidas I, Kalomenidis I, Porcel JM, Robinson BW, Stathopoulos GT. Malignant pleural effusion: from bench to bedside. Eur Respir Rev. 2016 Jun;25(140):189-98. doi: 10.1183/16000617.0019-2016. PMID 27246596
- [Background] Antony VB, Loddenkemper R, Astoul P, Boutin C, Goldstraw P, Hott J, Rodriguez Panadero F, Sahn SA. Management of malignant pleural effusions. Eur Respir J. 2001 Aug;18(2):402-19. doi: 10.1183/09031936.01.00225601. No abstract available. PMID 11529302
- [Background] Chernow B, Sahn SA. Carcinomatous involvement of the pleura: an analysis of 96 patients. Am J Med. 1977 Nov;63(5):695-702. doi: 10.1016/0002-9343(77)90154-1. No abstract available. PMID 930945